CLINICAL TRIAL: NCT04084769
Title: Immunogenicity and Safety of a Booster Dose of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Adolescents and Adults
Brief Title: Study to Evaluate the Immune Response After a Booster Dose of a Quadrivalent Meningococcal (MenACYW) Conjugate Vaccine When Administered Alone or Concomitantly With a Licensed Meningococcal Serogroup B Vaccine, in Participants Who Received Primary Quadrivalent Meningococcal Conjugate Vaccine (MCV4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MET59; U1111-1217-2137 (Other: UTN); 2019-004461-41 (EudraCT Number)
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Results first posted 2021-08-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Meningococcal Immunisation (Healthy Volunteers)
MeSH Terms: interventions — 4CMenB vaccine; MenB-FHbp vaccine

STUDY DESIGN:
Intervention Model Description: Partially-randomized design: all participants primed with MenACYW Conjugate vaccine who meet the inclusion/exclusion criteria were randomly assigned to Group 1, 3, or 4, while participants primed with Menveo vaccine were automatically allocated to Group 2 (not randomized).
Masking Description: The laboratory personnel who performed the serology testing were blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1: MenACYW Conjugate vaccine (Experimental): Participants who received a single dose of MenACYW Conjugate vaccine in previous studies MET50 (NCT02199691) or MET43 (NCT02842853), received a single intramuscular (IM) dose of MenACYW Conjugate vaccine, at Day 0 in the present study (MET59).
  Interventions: Biological: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid Conjugate vaccine MenACYW Conjugate vaccine
- Group 2: MenACYW Conjugate vaccine (Menveo Vaccine-primed) (Experimental): Participants who received a single dose of Menveo vaccine in previous study MET50 or outside of Sanofi Pasteur trials, received a single IM dose of MenACYW Conjugate vaccine, at Day 0 in the present study (MET59).
  Interventions: Biological: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid Conjugate vaccine MenACYW Conjugate vaccine
- Group 3: MenACYW Conjugate vaccine + Trumenba vaccine (Experimental): Participants who received a single dose of MenACYW Conjugate vaccine in previous studies MET50 or MET43, received a single IM dose of MenACYW Conjugate vaccine, concomitantly with 1 dose of Trumenba vaccine at Day 0 in the present study (MET59).
  Interventions: Biological: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid Conjugate vaccine MenACYW Conjugate vaccine; Biological: Meningococcal Group B vaccine (Trumenba®)
- Group 4: MenACYW Conjugate vaccine + Bexsero vaccine (Experimental): Participants who received a single dose of MenACYW Conjugate vaccine in previous studies MET50 or MET43, received a single IM dose of MenACYW Conjugate vaccine, concomitantly with 1 dose of Bexsero vaccine at Day 0 in the present study (MET59).
  Interventions: Biological: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid Conjugate vaccine MenACYW Conjugate vaccine; Biological: Meningococcal group B vaccine (Bexsero®)

INTERVENTIONS:
Biological: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid Conjugate vaccine MenACYW Conjugate vaccine — Pharmaceutical form: Solution for injection Route of administration: IM
Biological: Meningococcal Group B vaccine (Trumenba®) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: IM
  Other Names: Trumenba®
  Arms: Group 3: MenACYW Conjugate vaccine + Trumenba vaccine
Biological: Meningococcal group B vaccine (Bexsero®) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: IM
  Other Names: Bexsero®
  Arms: Group 4: MenACYW Conjugate vaccine + Bexsero vaccine

SUMMARY:
Primary Objective:

To demonstrate the vaccine seroresponse sufficiency of meningococcal serogroups A, C, Y, and W following the administration of a booster dose of meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine:

* In Group 1 participants who were first vaccinated with 1 dose of MenACYW Conjugate vaccine 3-6 years before the booster dose.
* In Group 2 participants who were first vaccinated with 1 dose of Menveo vaccine (meningococcal [Groups A, C, Y and W135] Oligosaccharide Diphtheria CRM197 Conjugate vaccine) 3-6 years before the booster dose.

Secondary Objective:

To describe:

* The vaccine seroresponse, seroprotection (serum bactericidal assay using human complement [hSBA] titer greater than or equal to [>=]1:8), and antibody responses (geometric mean titers [GMTs]) of meningococcal serogroups A, C, Y, and W measured using hSBA in serum specimens collected 6 days (±1 day) after vaccination in a subset of 50 participants per group (Groups 1 and 2).
* The vaccine seroresponse, seroprotection (hSBA titer >=1:8), and antibody responses (GMTs) to serogroups A, C, Y, and W measured using hSBA on Day (D)0 (pre-vaccination) and D30 (+14 days) after vaccination with MenACYW Conjugate vaccine alone (Groups 1 and 2).
* The antibody persistence (GMTs and vaccine seroprotection; hSBA titer >=1:8) of meningococcal serogroups A, C, Y, and W before a booster dose in participants who received either MenACYW Conjugate vaccine or Menveo vaccine 3-6 years earlier.
* The antibody persistence (GMTs and vaccine seroprotection; hSBA titer >=1:8) of meningococcal serogroups A, C, Y, and W in participants who received either a single dose MenACYW Conjugate vaccine (participants randomized to MET59 Groups 1, 3, and 4) or Menveo vaccine (participants assigned to MET59 Group 2), as part of study MET50, or MET43 (participants randomized to MET59 Groups 1, 3 and 4).
* To describe the vaccine seroresponse, seroprotection (hSBA titer >=1:8), and antibody responses (GMTs) to the antigens present in MenACYW Conjugate vaccine, when MenACYW Conjugate vaccine was given concomitantly with meningococcal serogroup B (MenB) vaccine (Groups 3 and 4), compared to those when it was given alone (Group 1).

DETAILED DESCRIPTION:
Study duration per participant was approximately 6 months including: 1 day of screening and vaccination, 1 or 2 additional visits at Day 6 and Day 30, 2 phone calls and a safety follow-up/end of study visit, at Day 8 and Day 180 after vaccine administration, respectively.

Safety assessment included solicited reactions within 7 days after vaccination, unsolicited adverse events (AEs) up to 30 days after vaccination, serious adverse events (SAEs) throughout the study.

ELIGIBILITY:
Inclusion criteria :

* Aged >= 13 to less than (<) 26 years on the day of inclusion.
* Participants participated in and completed study MET50 (MET50 Groups 1, 2, or 3 only) or study MET43 (MET43 Groups 1, 2, or 3 only).
* For MET59 Group 2 only (Menveo vaccine-primed participants only; enrichment population): participants had a documented record of having received 1 dose of Menveo vaccine 3-6 years earlier either as part of a clinical trial or as routine vaccination. Participants who participated in MET50 Group 4 can be enrolled if they fulfill this criterion.
* Participants aged 13 to < 18 years: assent form had been signed and dated by the participant and informed consent form (ICF) had been signed and dated by the parent or guardian.
* Participants aged >=18 (or legal age of majority, if different from 18 years of age) to < 26 years: ICF had been signed and dated by the participants.
* Participant aged 13 to < 18 years: both the participant and parent or guardian were able to attend all scheduled visits and complied with all trial procedures.
* Participants aged >=18 (or legal age of majority, if different from 18 years of age) to < 26 years: able to attend all scheduled visits and complied with all trial procedures.

Exclusion criteria:

* Participant was pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination. To be considered of non-childbearing potential, a female must be pre-menarche, or post-menopausal for at least 1 year, or surgically sterile.
* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine before Visit 3 (Day 30) except for influenza vaccination, which might be received at least 2 weeks before study investigational vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Receipt of any meningococcal vaccine including a licensed or investigational MenACWY vaccine or MenB vaccine since participation in study MET50 or MET43.
* Menveo vaccine-primed participants only (enrichment group for Group 2): receipt of more than 1 dose of Menveo vaccine or vaccination with another licensed or investigational MenACWY vaccine or with a licensed or investigational MenB vaccine.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial (specifically but not limited to participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Personal history of Guillain-Barré syndrome.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine within at least 10 years of the proposed study vaccination.
* Verbal report of thrombocytopenia, contraindicating IM vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
* Current alcohol abuse or drug addiction.
* Chronic illness (e.g., Human immunodeficiency viruses, hepatitis B, hepatitis C) that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >= 100.4 degree Fahrenheit). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 13 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 570 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (30):
- United States (29):
  - Investigational Site Number 8400012, Birmingham, Alabama
  - Investigational Site Number 8400005, San Diego, California
  - Investigational Site Number 8400013, Bardstown, Kentucky
  - Investigational Site Number 8400033, Lexington, Kentucky
  - Investigational Site Number 8400034, Bridgeton, Missouri
  - Investigational Site Number 8400027, Lincoln, Nebraska
  - Investigational Site Number 8400002, Lincoln, Nebraska
  - Investigational Site Number 8400004, Lincoln, Nebraska
  - Investigational Site Number 8400030, Dayton, Ohio
  - Investigational Site Number 8400028, South Euclid, Ohio
  - Investigational Site Number 8400009, Norman, Oklahoma
  - Investigational Site Number 8400038, Erie, Pennsylvania
  - Investigational Site Number 8400039, Charleston, South Carolina
  - Investigational Site Number 8400018, Kingsport, Tennessee
  - Investigational Site Number 8400029, Tullahoma, Tennessee
  - Investigational Site Number 8400031, Kaysville, Utah
  - Investigational Site Number 8400001, Layton, Utah
  - Investigational Site Number 8400014, Layton, Utah
  - Investigational Site Number 8400040, Orem, Utah
  - Investigational Site Number 8400011, Provo, Utah
  - Investigational Site Number 8400023, Roy, Utah
  - Investigational Site Number 8400003, Salt Lake City, Utah
  - Investigational Site Number 8400007, Salt Lake City, Utah
  - Investigational Site Number 8400022, Salt Lake City, Utah
  - Investigational Site Number 8400015, South Jordan, Utah
  - Investigational Site Number 8400036, South Jordan, Utah
  - Investigational Site Number 8400032, Syracuse, Utah
  - Investigational Site Number 8400024, West Jordan, Utah
  - Investigational Site Number 8400037, Charlottesville, Virginia
- Investigational Site Number 6300001, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Zambrano B, Peterson J, Deseda C, Julien K, Spiegel CA, Seyler C, Simon M, Hoki R, Anderson M, Brabec B, Anez G, Shi J, Pan J, Hagenbach A, Von Barbier D, Varghese K, Jordanov E, Dhingra MS. Quadrivalent meningococcal tetanus toxoid-conjugate booster vaccination in adolescents and adults: phase III randomized study. Pediatr Res. 2023 Sep;94(3):1035-1043. doi: 10.1038/s41390-023-02478-5. Epub 2023 Mar 10. PMID 36899125
- See also: MET59 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25314&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 03-September-2019 to 07-March-2020 at 30 active sites in the United States and Puerto Rico.
Pre-assignment Details: A total of 570 participants who received meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine or Menveo (meningococcal Group B) vaccine either in Study MET50 (NCT02199691), or Study MET43 (NCT02842853), or outside of Sanofi Pasteur trials were enrolled in the present study (MET59).
Groups:
- Group 1: MenACYW Conjugate Vaccine: Participants who received a single dose of MenACYW Conjugate vaccine in previous studies MET50 or MET43, received a single intramuscular (IM) dose of MenACYW Conjugate vaccine, at Day 0 in the present study (MET59).
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed) | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine
Started | 191 | 190 | 95 | 94
Safety Analysis Set (SAfAS) (Participants who had received at least one dose of study vaccine in MET59 and had available safety data.) | 186 | 184 | 93 | 92
Full Analysis Set (Participants who had a valid pre-vaccination serology result.) | 191 | 190 | 95 | 94
Per-Protocol Analysis Set 1 (PPAS1) (Participants who received at least 1 dose of the study vaccine in MET59 and had a valid post-vaccination serology result with no relevant protocol deviation; defined for evaluating the immune response of MenACYW vaccine measured by serum bactericidal assay using human complement (hSBA) assessed at Day 06 after vaccination in Groups 1 and 2.) | 46 | 45 | 0 | 0
Per-Protocol Analysis Set 2 (PPAS2) (Participants who received at least 1 dose of the study vaccine in MET59 and had a valid post-vaccination serology result with no relevant protocol deviation; defined for evaluating the immune response of MenACYW vaccine measured by hSBA or serum bactericidal assay using baby rabbit complement (rSBA) assessed at Day 30 after vaccination.) | 174 | 176 | 90 | 89
Completed | 187 | 186 | 95 | 92
Not Completed | 4 | 4 | 0 | 2
Not completed — Protocol Violation | 1 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Withdrawal by parent/guardian | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Participants who received a single dose of MenACYW Conjugate vaccine in previous studies MET50 or MET43, received a single IM dose of MenACYW Conjugate vaccine, at Day 0 in the present study (MET59).
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed) | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine | Total
Number analyzed (Participants) | 191 | 190 | 95 | 94 | 570
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.59) | 15.8 (1.37) | 15.1 (1.12) | 15.3 (1.34) | 15.4 (1.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 85 | 41 | 45 | 270
  Male | 92 | 105 | 54 | 49 | 300
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 2
  Black or African American | 19 | 16 | 7 | 7 | 49
  White | 163 | 165 | 83 | 86 | 497
  More than one race | 8 | 6 | 5 | 0 | 19
  Unknown or Not Reported | 0 | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Vaccine Seroresponse Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by Serum Bactericidal Assay Using Human Complement (hSBA). The hSBA vaccine seroresponse was defined as a post-vaccination hSBA titer greater than or equal to (>=) 1:16 for participants with pre-vaccination hSBA titer less than (<) 1:8, or a >= 4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >= 1:8. Immune response was considered sufficient if lower limit of the 1-sided 97.5% CI for percentage of participants with hSBA seroresponse against serogroups A, C, Y and W was greater than 75%.
Time Frame: Day 30 (post-vaccination) in study MET59
Population: Analysis was performed on Per-Protocol Analysis Set 2 (PPAS2) population that included participants who received 1 dose of study vaccine in MET59 and had a valid post-vaccination serology result with no relevant protocol deviation; defined for evaluating the immune response of MenACYW vaccine measured by hSBA or rSBA assessed at Day 30 after vaccination. For this outcome measure, data were not planned to be collected and analyzed for Groups 3, and 4 as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine
Number analyzed (Participants) | 174
percentage of participants
  Serogroup A | 94.8 [90.4 to 97.6]
  Serogroup C | 97.1 [93.4 to 99.1]
  Serogroup Y | 98.9 [95.9 to 99.9]
  Serogroup W | 97.7 [94.2 to 99.4]

2. Primary Outcome: Percentage of Participants With Vaccine Seroresponse Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 2
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. The hSBA vaccine seroresponse was defined as a post-vaccination hSBA titer >=1:16 for participants with pre-vaccination hSBA titer <1:8, or a >=4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >=1:8. Immune response was considered sufficient if lower limit of the 1-sided 97.5% CI for percentage of participants with hSBA seroresponse against serogroups A, C, Y and W was greater than 75%.
Time Frame: Day 30 (post-vaccination) in study MET59
Population: Analysis was performed on PPAS2 population. For this outcome measure, data were not planned to be collected and analyzed for Groups 3, and 4 as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed)
Number analyzed (Participants) | 176
percentage of participants
  Serogroup A | 93.2 [88.4 to 96.4]
  Serogroup C | 98.9 [96.0 to 99.9]
  Serogroup Y | 100 [97.9 to 100]
  Serogroup W | 98.9 [96.0 to 99.9]

3. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1 and 2
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. The hSBA vaccine seroresponse was defined as a post-vaccination hSBA titer >=1:16 for participants with pre-vaccination hSBA titer <1:8, or a >=4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >=1:8.
Time Frame: Day 6 (post-vaccination) in study MET59
Population: Analysis was performed on Per-Protocol Analysis Set 1 (PPAS1) population that included participants who received 1 dose of study vaccine in MET59 and had valid serology result with no relevant protocol deviations; defined for evaluating the immune response of MenACYW vaccine measured by hSBA assessed at Day 06 after vaccination in Groups 1 and 2. For this outcome measure, data were not planned to be collected and analyzed for Groups 3, and 4 as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed)
Number analyzed (Participants) | 46 | 45
percentage of participants
  Serogroup A | 82.6 [68.6 to 92.2] | 77.8 [62.9 to 88.8]
  Serogroup C | 89.1 [76.4 to 96.4] | 93.3 [81.7 to 98.6]
  Serogroup Y | 95.7 [85.2 to 99.5] | 91.1 [78.8 to 97.5]
  Serogroup W | 97.8 [88.5 to 99.9] | 88.9 [75.9 to 96.3]

4. Secondary Outcome: Percentage of Participants With Vaccine Seroprotection Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1 and 2
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. Seroprotection was defined as hSBA titer >=1:8.
Time Frame: Day 6 (post-vaccination) in study MET59
Population: Analysis was performed on PPAS1 population. For this outcome measure, data were not planned to be collected and analyzed for Groups 3, and 4 as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed)
Number analyzed (Participants) | 46 | 45
percentage of participants
  Serogroup A | 91.3 [79.2 to 97.6] | 95.6 [84.9 to 99.5]
  Serogroup C | 100 [92.3 to 100] | 97.8 [88.2 to 99.9]
  Serogroup Y | 97.8 [88.5 to 99.9] | 100 [92.1 to 100]
  Serogroup W | 100 [92.3 to 100] | 100 [92.1 to 100]

5. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1 and 2
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 6 (post-vaccination) in study MET59
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed)
Number analyzed (Participants) | 46 | 45
titers
  Serogroup A | 289 [133 to 625] | 161 [93.0 to 280]
  Serogroup C | 3799 [2504 to 5763] | 919 [500 to 1690]
  Serogroup Y | 1658 [973 to 2826] | 800 [467 to 1371]
  Serogroup W | 1928 [1187 to 3131] | 708 [463 to 1082]

6. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1 and 2
Description: as for outcome 3
Time Frame: Day 30 (post-vaccination) in study MET59
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed)
Number analyzed (Participants) | 174 | 176
percentage of participants
  Serogroup A | 94.8 [90.4 to 97.6] | 93.2 [88.4 to 96.4]
  Serogroup C | 97.1 [93.4 to 99.1] | 98.9 [96.0 to 99.9]
  Serogroup Y | 98.9 [95.9 to 99.9] | 100 [97.9 to 100]
  Serogroup W | 97.7 [94.2 to 99.4] | 98.9 [96.0 to 99.9]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed); Serogroup A; Test type: Other — 95% Confidence Interval (CI) of the difference in percentage was calculated from the Wilson Score method without continuity correction; Difference in percentage = 1.65, 95% CI 2-sided [-3.58 to 6.95]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed); Serogroup C; Test type: Other — 95% CI of the difference in percentage was calculated from the Wilson Score Method without continuity correction; Difference in percentage = -1.74, 95% CI 2-sided [-5.50 to 1.60]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed); Serogroup Y; Test type: Other — 95% CI of the difference in percentage was calculated from the Wilson Score Method without continuity correction; Difference in percentage = -1.15, 95% CI 2-sided [-4.09 to 1.14]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed); Serogroup W; Test type: Other — 95% CI of the difference in percentage was calculated from the Wilson Score Method without continuity correction; Difference in percentage = -1.16, 95% CI 2-sided [-4.72 to 2.07]

7. Secondary Outcome: Percentage of Participants With Vaccine Seroprotection Against Meningococcal Serogroups A, C, Y, and W at Day 0 and at Day 30 Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1 and 2
Description: Antibody titers against meningococcal serogroups A, C, W, and Y were measured by hSBA. Seroprotection were defined as hSBA titer >=1:8.
Time Frame: Day 0 (pre-vaccination) and Day 30 (post-vaccination) in study MET59
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed)
Number analyzed (Participants) | 174 | 176
percentage of participants
  Serogroup A: Day 0 | 71.3 [63.9 to 77.9] | 71.0 [63.7 to 77.6]
  Serogroup A: Day 30 | 99.4 [96.8 to 100] | 99.4 [96.9 to 100]
  Serogroup C: Day 0 | 87.9 [82.1 to 92.4] | 50.6 [42.9 to 58.2]
  Serogroup C: Day 30 | 100 [97.9 to 100] | 100 [97.9 to 100]
  Serogroup Y: Day 0 | 79.9 [73.2 to 85.6] | 52.8 [45.2 to 60.4]
  Serogroup Y: Day 30 | 100 [97.9 to 100] | 100 [97.9 to 100]
  Serogroup W: Day 0 | 86.2 [80.2 to 91.0] | 77.8 [71.0 to 83.7]
  Serogroup W: Day 30 | 100 [97.9 to 100] | 100 [97.9 to 100]

8. Secondary Outcome: GMTs of Antibodies Against Meningococcal Serogroups A, C, Y, and W at Day 0 and at Day 30 Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1 and 2
Description: as for outcome 5
Time Frame: Day 0 (pre-vaccination) and Day 30 (post-vaccination) in study MET59
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed)
Number analyzed (Participants) | 174 | 176
titers
  Serogroup A: Day 0 | 11.7 [9.89 to 13.8] | 11.5 [9.72 to 13.7]
  Serogroup A: Day 30 | 502 [388 to 649] | 399 [318 to 502]
  Serogroup C: Day 0 | 36.6 [28.8 to 46.7] | 10.2 [8.03 to 13.0]
  Serogroup C: Day 30 | 3708 [3146 to 4369] | 2533 [2076 to 3091]
  Serogroup Y: Day 0 | 20.5 [16.6 to 25.2] | 8.35 [6.70 to 10.4]
  Serogroup Y: Day 30 | 2308 [1925 to 2767] | 3036 [2547 to 3620]
  Serogroup W: Day 0 | 27.0 [22.0 to 33.1] | 14.8 [12.2 to 18.1]
  Serogroup W: Day 30 | 2290 [1934 to 2711] | 2574 [2178 to 3041]

9. Secondary Outcome: Percentage of Participants With Vaccine Seroprotection Against Meningococcal Serogroups A, C, Y, and W at Day 0
Description: as for outcome 4
Time Frame: Day 0 (pre-vaccination) in study MET59
Population: Analysis was performed on full analysis set which included all participants who had a valid pre-vaccination serology result. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed) | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine
Number analyzed (Participants) | 191 | 190 | 95 | 94
percentage of participants
  Serogroup A: number analyzed (Participants) | 191 | 190 | 95 | 93
  Serogroup A | 72.3 [65.3 to 78.5] | 71.1 [64.0 to 77.4] | 73.7 [63.6 to 82.2] | 73.1 [62.9 to 81.8]
  Serogroup C | 86.9 [81.3 to 91.3] | 52.6 [45.3 to 59.9] | 86.3 [77.7 to 92.5] | 85.1 [76.3 to 91.6]
  Serogroup Y: number analyzed (Participants) | 191 | 190 | 94 | 94
  Serogroup Y | 79.1 [72.6 to 84.6] | 55.3 [47.9 to 62.5] | 88.3 [80.0 to 94.0] | 80.9 [71.4 to 88.2]
  Serogroup W: number analyzed (Participants) | 191 | 190 | 95 | 93
  Serogroup W | 86.9 [81.3 to 91.3] | 77.9 [71.3 to 83.6] | 90.5 [82.8 to 95.6] | 91.4 [83.8 to 96.2]

10. Secondary Outcome: GMTs of Antibodies Against Meningococcal Serogroups A, C, Y, and W at Day 0
Description: as for outcome 5
Time Frame: Day 0 (pre-vaccination) in study MET59
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed) | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine
Number analyzed (Participants) | 191 | 190 | 95 | 94
titers
  Serogroup A: number analyzed (Participants) | 191 | 190 | 95 | 93
  Serogroup A | 12.3 [10.5 to 14.5] | 12.2 [10.2 to 14.6] | 12.8 [10.0 to 16.3] | 12.7 [9.70 to 16.6]
  Serogroup C | 34.5 [27.4 to 43.6] | 11.9 [9.17 to 15.3] | 38.4 [27.3 to 54.0] | 43.3 [29.8 to 63.0]
  Serogroup Y: number analyzed (Participants) | 191 | 190 | 94 | 94
  Serogroup Y | 19.8 [16.2 to 24.2] | 9.19 [7.39 to 11.4] | 26.0 [19.6 to 34.5] | 22.0 [16.1 to 30.0]
  Serogroup W: number analyzed (Participants) | 191 | 190 | 95 | 93
  Serogroup W | 27.4 [22.4 to 33.4] | 15.1 [12.5 to 18.3] | 28.1 [21.8 to 36.2] | 32.7 [24.5 to 43.7]

11. Secondary Outcome: Percentage of Participants Achieving Vaccine Seroprotection Against Meningococcal Serogroups A, C, Y, and W at Day 0 and 30 Days Post-Vaccination in Study MET50 or MET43
Description: as for outcome 4
Time Frame: Day 0 (pre-vaccination), Day 30 (post-vaccination) in study MET50 or MET43
Population: Analysis was performed on full analysis set which included all participants who had a valid pre-vaccination serology result. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category. For this outcome measure, data were planned to be collected and analyzed for pooled population of groups 1, 3 and 4 as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pooled Groups 1, 3 and 4: MenACYW Conjugate Vaccine: Included all participants of Groups 1, 3 and 4 who received MenACYW Conjugate vaccine in previous studies MET50 or MET43. Participants of Group 1 participants received a single IM dose of MenACYW Conjugate vaccine and Group 3 and 4 participants received a single IM dose of MenACYW Conjugate vaccine, concomitantly with 1 dose of Trumenba vaccine and Bexsero vaccine, respectively, at Day 0 in the present study (MET59).
Arm/Group | Pooled Groups 1, 3 and 4: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed)
Number analyzed (Participants) | 376 | 134
percentage of participants
  Serogroup A: Day 0 of MET50 or MET43 | 54.5 [49.3 to 59.6] | 35.8 [27.7 to 44.6]
  Serogroup A: Day 30 of MET50 or MET43: number analyzed (Participants) | 376 | 133
  Serogroup A: Day 30 of MET50 or MET43 | 94.7 [91.9 to 96.7] | 81.2 [73.5 to 87.5]
  Serogroup C: Day 0 of MET50 or MET43 | 18.6 [14.8 to 22.9] | 12.7 [7.6 to 19.5]
  Serogroup C: Day 30 of MET50 or MET43: number analyzed (Participants) | 376 | 132
  Serogroup C: Day 30 of MET50 or MET43 | 98.1 [96.2 to 99.2] | 74.2 [65.9 to 81.5]
  Serogroup Y: Day 0 of MET50 or MET43 | 4.5 [2.7 to 7.1] | 3.7 [1.2 to 8.5]
  Serogroup Y: Day 30 of MET50 or MET43: number analyzed (Participants) | 376 | 133
  Serogroup Y: Day 30 of MET50 or MET43 | 97.9 [95.9 to 99.1] | 88.7 [82.1 to 93.5]
  Serogroup W: Day 0 of MET50 or MET43 | 39.9 [34.9 to 45.0] | 40.3 [31.9 to 49.1]
  Serogroup W: Day 30 of MET50 or MET43: number analyzed (Participants) | 376 | 133
  Serogroup W: Day 30 of MET50 or MET43 | 100 [99.0 to 100] | 93.2 [87.5 to 96.9]

12. Secondary Outcome: GMTs of Antibodies Against Meningococcal Serogroups A, C, Y, and W at Day 0 and 30 Days Post Vaccination in Either Study MET50 or MET43 and Pre Vaccination in Study MET59
Description: as for outcome 5
Time Frame: Day 0 (pre-vaccination) and Day 30 (post-vaccination) in study MET50 or MET43; Day 0 (pre-vaccination) in study MET59
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Pooled Groups 1, 3 and 4: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed)
Number analyzed (Participants) | 380 | 140
titers
  Serogroup A: Day 0 of MET50 or MET43: number analyzed (Participants) | 376 | 134
  Serogroup A: Day 0 of MET50 or MET43 | 7.28 [6.53 to 8.11] | 5.72 [4.75 to 6.87]
  Serogroup A: Day 30 of MET50 or MET43: number analyzed (Participants) | 376 | 133
  Serogroup A: Day 30 of MET50 or MET43 | 45.2 [39.9 to 51.1] | 32.8 [25.0 to 43.1]
  Serogroup A: Day 0 of MET59: number analyzed (Participants) | 379 | 140
  Serogroup A: Day 0 of MET59 | 12.5 [11.1 to 14.1] | 11.6 [9.41 to 14.3]
  Serogroup C: Day 0 of MET50 or MET43: number analyzed (Participants) | 376 | 134
  Serogroup C: Day 0 of MET50 or MET43 | 3.48 [3.22 to 3.76] | 2.98 [2.69 to 3.30]
  Serogroup C: Day 30 of MET50 or MET43: number analyzed (Participants) | 376 | 132
  Serogroup C: Day 30 of MET50 or MET43 | 417 [348 to 500] | 49.7 [32.4 to 76.4]
  Serogroup C: Day 0 of MET59 | 37.5 [31.6 to 44.5] | 11.0 [8.09 to 14.9]
  Serogroup Y: Day 0 of MET50 or MET43: number analyzed (Participants) | 376 | 134
  Serogroup Y: Day 0 of MET50 or MET43 | 2.36 [2.22 to 2.50] | 2.30 [2.13 to 2.48]
  Serogroup Y: Day 30 of MET50 or MET43: number analyzed (Participants) | 376 | 133
  Serogroup Y: Day 30 of MET50 or MET43 | 91.0 [78.6 to 105] | 36.1 [27.2 to 47.8]
  Serogroup Y: Day 0 of MET59: number analyzed (Participants) | 379 | 140
  Serogroup Y: Day 0 of MET59 | 21.8 [18.8 to 25.1] | 8.49 [6.50 to 11.1]
  Serogroup W: Day 0 of MET50 or MET43: number analyzed (Participants) | 376 | 134
  Serogroup W: Day 0 of MET50 or MET43 | 5.34 [4.76 to 6.00] | 5.54 [4.57 to 6.72]
  Serogroup W: Day 30 of MET50 or MET43: number analyzed (Participants) | 376 | 133
  Serogroup W: Day 30 of MET50 or MET43 | 82.7 [73.6 to 92.9] | 45.1 [34.3 to 59.4]
  Serogroup W: Day 0 of MET59: number analyzed (Participants) | 379 | 140
  Serogroup W: Day 0 of MET59 | 28.8 [25.1 to 33.0] | 14.9 [11.9 to 18.6]

13. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1, 3 and 4
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. The hSBA vaccine seroresponse was defined as a post-vaccination hSBA titer >=1:16 for participants with pre-vaccination hSBA titer <1:8, or a >= 4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >=1:8.
Time Frame: Day 30 (post-vaccination) in study MET59
Population: Analysis was performed on PPAS2 population. Here, 'number analyzed' = participants with available data for each specified category. For this outcome measure, data were planned to be collected and analyzed for individual groups 1, 3 and 4 and for pooled population of groups 3 and 4 only, and not for group 2 as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pooled Groups 3 and 4: MenACYW Conjugate Vaccine: Included all participants of Groups 3 and 4 who received MenACYW Conjugate vaccine in previous studies MET50 or MET43. Participants of Group 3 and 4 participants received a single IM dose of MenACYW Conjugate vaccine, concomitantly with 1 dose of Trumenba vaccine and Bexsero vaccine at Day 0 in the present study (MET59).
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine | Pooled Groups 3 and 4: MenACYW Conjugate Vaccine
Number analyzed (Participants) | 174 | 90 | 89 | 179
percentage of participants
  Serogroup A: number analyzed (Participants) | 174 | 90 | 88 | 178
  Serogroup A | 94.8 [90.4 to 97.6] | 93.3 [86.1 to 97.5] | 95.5 [88.8 to 98.7] | 94.4 [89.9 to 97.3]
  Serogroup C: number analyzed (Participants) | 174 | 90 | 88 | 178
  Serogroup C | 97.1 [93.4 to 99.1] | 97.8 [92.2 to 99.7] | 96.6 [90.4 to 99.3] | 97.2 [93.6 to 99.1]
  Serogroup Y: number analyzed (Participants) | 174 | 89 | 89 | 178
  Serogroup Y | 98.9 [95.9 to 99.9] | 98.9 [93.9 to 100] | 97.8 [92.1 to 99.7] | 98.3 [95.2 to 99.7]
  Serogroup W: number analyzed (Participants) | 174 | 90 | 88 | 178
  Serogroup W | 97.7 [94.2 to 99.4] | 98.9 [94.0 to 100] | 96.6 [90.4 to 99.3] | 97.8 [94.3 to 99.4]

14. Secondary Outcome: Percentage of Participants With Vaccine Seroprotection Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1, 3 and 4
Description: as for outcome 4
Time Frame: Day 0 (pre-vaccination) and Day 30 (post-vaccination) in study MET59
Population: Analysis was performed on PPAS2 population. Here, 'number analyzed'=participants with available data for each specified category. For this outcome measure, data were planned to be collected and analyzed for individual groups 1, 3 and 4 and for pooled population of groups 3 and 4 only, and not for group 2 as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine | Pooled Groups 3 and 4: MenACYW Conjugate Vaccine
Number analyzed (Participants) | 174 | 90 | 89 | 179
percentage of participants
  Serogroup A: Day 0: number analyzed (Participants) | 174 | 90 | 88 | 178
  Serogroup A: Day 0 | 71.3 [63.9 to 77.9] | 73.3 [63.0 to 82.1] | 71.6 [61.0 to 80.7] | 72.5 [65.3 to 78.9]
  Serogroup A: Day 30 | 99.4 [96.8 to 100] | 98.9 [94.0 to 100] | 100 [95.9 to 100] | 99.4 [96.9 to 100]
  Serogroup C: Day 0 | 87.9 [82.1 to 92.4] | 86.7 [77.9 to 92.9] | 86.5 [77.6 to 92.8] | 86.6 [80.7 to 91.2]
  Serogroup C: Day 30: number analyzed (Participants) | 174 | 90 | 88 | 178
  Serogroup C: Day 30 | 100 [97.9 to 100] | 100 [96.0 to 100] | 100 [95.9 to 100] | 100 [97.9 to 100]
  Serogroup Y: Day 0: number analyzed (Participants) | 174 | 89 | 89 | 178
  Serogroup Y: Day 0 | 79.9 [73.2 to 85.6] | 89.9 [81.7 to 95.3] | 80.9 [71.2 to 88.5] | 85.4 [79.3 to 90.2]
  Serogroup Y: Day 30 | 100 [97.9 to 100] | 100 [96.0 to 100] | 100 [95.9 to 100] | 100 [98.0 to 100]
  Serogroup W: Day 0: number analyzed (Participants) | 174 | 90 | 88 | 178
  Serogroup W: Day 0 | 86.2 [80.2 to 91.0] | 91.1 [83.2 to 96.1] | 90.9 [82.9 to 96.0] | 91.0 [85.8 to 94.8]
  Serogroup W: Day 30 | 100 [97.9 to 100] | 100 [96.0 to 100] | 100 [95.9 to 100] | 100 [98.0 to 100]

15. Secondary Outcome: GMTs of Antibodies Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine in Study MET59: Group 1, 3 and 4
Description: as for outcome 5
Time Frame: Day 0 (pre-vaccination) and Day 30 (post-vaccination) in study MET59
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine | Pooled Groups 3 and 4: MenACYW Conjugate Vaccine
Number analyzed (Participants) | 174 | 90 | 89 | 179
titers
  Serogroup A: Day 0: number analyzed (Participants) | 174 | 90 | 88 | 178
  Serogroup A: Day 0 | 11.7 [9.89 to 13.8] | 12.5 [9.78 to 16.0] | 12.3 [9.37 to 16.2] | 12.4 [10.4 to 14.9]
  Serogroup A: Day 30 | 502 [388 to 649] | 593 [426 to 825] | 667 [477 to 933] | 629 [498 to 794]
  Serogroup C: Day 0 | 36.6 [28.8 to 46.7] | 37.6 [26.6 to 53.3] | 42.4 [29.4 to 61.0] | 39.9 [31.1 to 51.2]
  Serogroup C: Day 30: number analyzed (Participants) | 174 | 90 | 88 | 178
  Serogroup C: Day 30 | 3708 [3146 to 4369] | 4741 [3882 to 5791] | 3472 [2667 to 4518] | 4064 [3446 to 4793]
  Serogroup Y: Day 0: number analyzed (Participants) | 174 | 89 | 89 | 178
  Serogroup Y: Day 0 | 20.5 [16.6 to 25.2] | 25.5 [19.4 to 33.6] | 21.0 [15.4 to 28.7] | 23.2 [18.9 to 28.5]
  Serogroup Y: Day 30 | 2308 [1925 to 2767] | 2600 [2042 to 3311] | 2469 [1881 to 3241] | 2534 [2117 to 3034]
  Serogroup W: Day 0: number analyzed (Participants) | 174 | 90 | 88 | 178
  Serogroup W: Day 0 | 27.0 [22.0 to 33.1] | 28.3 [22.0 to 36.4] | 30.0 [22.5 to 40.1] | 29.1 [24.1 to 35.2]
  Serogroup W: Day 30 | 2290 [1934 to 2711] | 2702 [2134 to 3422] | 2064 [1601 to 2662] | 2363 [1988 to 2810]

ADVERSE EVENTS:
Time Frame: Unsolicited adverse event (AE) data were collected from Day 0 (pre-vaccination) up to Day 30 (post-vaccination) in MET59. The solicited reactions (SR) were collected within 7 days post-vaccination in MET59. Serious AEs data were collected up to 30 days post-vaccination in MET59.
Description: Analysis performed on SafAS population.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed) | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine
All-Cause Mortality (participants affected / at risk) | 0/186 | 0/184 | 0/93 | 0/92
Serious Adverse Events (participants affected / at risk) | 2/186 | 2/184 | 2/93 | 0/92
Other Adverse Events (participants affected / at risk) | 129/186 | 116/184 | 83/93 | 88/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=186) | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed) (N=184) | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine (N=93) | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine (N=92)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=186) | Group 2: MenACYW Conjugate Vaccine (Menveo Vaccine-primed) (N=184) | Group 3: MenACYW Conjugate Vaccine + Trumenba Vaccine (N=93) | Group 4: MenACYW Conjugate Vaccine + Bexsero Vaccine (N=92)
Injection Site Erythema (General disorders) | 12 (12) | 10 (10) | 15 (15) | 14 (19)
Injection Site Pain (General disorders) | 71 (71) | 63 (63) | 77 (114) | 85 (123)
Injection Site Swelling (General disorders) | 10 (10) | 3 (3) | 12 (13) | 15 (19)
Malaise (General disorders) | 50 (50) | 47 (47) | 36 (36) | 37 (37)
Nasopharyngitis (Infections and infestations) | 9 (10) | 6 (6) | 5 (5) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (10) | 8 (8) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 61 (61) | 64 (64) | 60 (61) | 58 (58)
Headache (Nervous system disorders) | 68 (69) | 67 (67) | 41 (42) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications

DOCUMENTS (2):
  • Study Protocol (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT04084769/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04084769/SAP_001.pdf